CLINICAL TRIAL: NCT07107204
Title: A Multicenter, Open-label, Single-arm Phase Ib/IIa Clinical Study to Evaluate the Safety and Efficacy of BT02 in Patients With Relapsed or Refractory Hematologic Malignancies
Brief Title: A Clinical Study of BT02 in Patients With Relapsed or Refractory Hematologic Malignancies
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biotroy Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BT02-201
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-07

CONDITIONS: Relapsed or Refractory Hematologic Malignancies; Leukemia; Lymphoma; Multiple Myeloma (MM)
MeSH Terms: conditions — Recurrence; Hematologic Neoplasms; Leukemia; Lymphoma; Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- dose escalation and expansion (Experimental)
  Interventions: Drug: BT02

INTERVENTIONS:
Drug: BT02 — BT02 monoclonal antibody injection with intravenous administration every 2 or 3 weeks

SUMMARY:
The goal of this clinical trial is to learn about the safety, tolerability and preliminary effectiveness of a treatment for patients with relapsed or refractory hematologic malignancies, regardless of gender, aged between 18(inclusive) and 70 years .

Participants will receive the investigational product intravenously every two or three weeks. The treatment will continue for a maximum of two years for those who do not show signs of disease progression or experience intolerable side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation with signed informed consent by the participant or their legal guardian and being willing and able to comply with all trial procedures.
2. Age:≥18 and <70 years, any gender.
3. Diagnosis:Confirmed hematologic malignancy (leukemia, lymphoma, or multiple myeloma) .
4. Leukemia-Specific Requirement:Bone marrow blast count ≥5% (morphological) at screening.
5. Measurable Disease.
6. Relapsed/Refractory Status.
7. Adequate organ and hematologic function.
8. An ECOG activity status score of 0-1.
9. A life expectancy of ≥ 3 months.
10. Eligible participants of childbearing potential (both males and females) must agree to using effective contraception throughout the study period.

Exclusion Criteria:

1. Acute promyelocytic leukemia (APL).
2. Patients with hereditary syndromes such as Fanconi anemia, Kostmann syndrome, Shwachman syndrome, or any other known bone marrow failure syndrome.
3. Patients with isolated extramedullary leukemia and multiple myeloma.
4. Patients with uncontrolled active central nervous system leukemia (CNSL).
5. Patients who have received anticancer therapy prior to administration.
6. A history of active autoimmune disease requiring systemic immunosuppressive therapy within the past 2 years.
7. A history of clinically significant cardiovascular disease, severe cardiac rhythm/conduction abnormalities ,severe pulmonary disease that may lead to severe episodes of dyspnea,head trauma, impaired consciousness, epilepsy, cerebral ischemia, or cerebral hemorrhagic disease.
8. A severe acute or chronic infection when enrollment.
9. Remaining the toxic reaction in previous anti-tumor therapy that has not recovered to ≤ Grade 1 .
10. Unresolved > grade 1 irAE or the history of a grade ≥ 3 irAE in previous immunotherapy, or known hypersensitivity to the formulation of the investigational product.
11. Patients undergoing acute graft-versus-host disease (GVHD) or moderate-to-severe chronic GVHD or systemic GVHD therapy.
12. A history of other type of malignancies.
13. Received a live attenuated vaccine within 28 days prior to the administration of the investigational product.
14. Poor compliance.
15. A history of alcohol/drugs abuse.
16. Current pregnancy or breastfeeding.
17. Other severe physical or mental illnesses or abnormal laboratory test results that the investigator deems unsuitable for participation in this study considering safety and compliance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Through the study completion, an average of 2.5 years
Dose limited toxicity(DLT) | Through the dose escalation phase, an average of 10 months
Maximum tolerable dose(MTD) | Through the dose escalation phase, an average of 10 months
Recommended phase 2 dose(RP2D) | Through the study completion, an average of 2.5 years

SECONDARY OUTCOMES:
Objective response rate (ORR) on tumor assessments | Through the study completion, an average of 2.5 years
Progression-free survival (PFS) on tumor assessments | Through the study completion, an average of 2.5 years
Overall survival (OS) | Through the study completion, an average of 2.5 years
Duration of response (DoR) on tumor assessments | Through the study completion, an average of 2.5 years
Disease control rate (DCR) on tumor assessments | Through the study completion, an average of 2.5years
Mean and median Area under the curve (AUC) of BT02 following first dose and repeated administration at each dose level | Through the study completion, an average of 2.5 years
Mean and median Maximum concentration (Cmax) of BT02 following first dose and repeated administration at each dose level | Through the study completion, an average of 2.5 years
ADA and NAb incidence | Through the study completion, an average of 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ying Wang, MD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences (IHCAMS)

IPD SHARING:
Plan to Share IPD: Undecided